CLINICAL TRIAL: NCT03617848
Title: Optimising Management of Patients With Heart Failure With Preserved Ejection Fraction in Primary Care
Acronym: OPTIMISEHFpEF
Status: Completed | Type: Observational
Sponsor: Professor Christi Deaton (Other)
Collaborators: University of Oxford (Other); Keele University (Other); University of Manchester (Other)
Responsible Party: Sponsor-Investigator, Professor Christi Deaton, Professor Christi Deaton, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: 234872
Record Dates: First submitted 2018-07-31; First posted 2018-08-07 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: HFpEF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma will be retained for future analysis as novel biomarkers emerge
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: A cohort of participants with suspected stable HFpEF will be recruited from the primary care setting. HFpEF diagnosis will be confirmed as per the 2016 European Society of Cardiology (ESC) guidelines for diagnosing HFpEF. All participants will undergo a series of assessments including but not limited to pulse wave velocity, 6 minute walk test, blood tests including natriuretic peptides (NT-Pro-BNP), ECG, physical assessments and a series of questionnaires. Those with confirmed HFpEF will be followed up at 6 and 12 months.

SUMMARY:
Heart failure (HF) accounts for 2% of National Health Service (NHS) expenditure, and 5% of emergency hospitalisations. Patients with HF with preserved ejection fraction (HFpEF) are older, have more comorbidities, have similarly poor or worse outcomes compared to patients with reduced ejection fraction (HFrEF), and currently lack an evidence base for treatment. The investigators hypothesise that outcomes of patients with HFpEF can be improved through optimised management and self-management of comorbidities, fluid status and lifestyle delivered in primary care in collaboration with specialists. The primary aim is to develop a programme of optimised management by improving understanding of needs and experiences of patients with HFpEF, clinical decision-making and management in primary care, and integrating research findings with patient and clinical expertise. The main objective for this work package is to identify patients with HFpEF in primary care and assess comorbidities and other factors, management, morbidity and mortality at one year. The methodology employed will be a longitudinal cohort study of 270 patients with HFpEF in primary care followed for 12 months.

DETAILED DESCRIPTION:
This work package of the study will use phenotyping and one-year follow-up of a community recruited cohort of patients with HFpEF or probable HFpEF to understand the characteristics and needs of this patient group. It involves a longitudinal cohort study conducted to identify patients with HFpEF in primary care and assess comorbidities, lifestyle factors, frailty, self-management, symptoms, quality of life, cognitive function, types of care received, management of risk factors and comorbidities, and one year morbidity and mortality. This will inform particular areas for assessment and management/self-management in the optimised programme. The investigators will also apply to NHS Digital who are the data controllers of Hospital Episode Statistics to check if participants have had any hospitals visits throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with diagnosed or suspected HFpEF (defined as: patients diagnosed with non-valvular HF that are i) not diagnosed with left ventricular systolic dysfunction or have a documented ejection fraction < 50%; or ii) do have a reported 'normal' or preserved EF, documented EF > 50%, or reported diastolic dysfunction without moderate to severe systolic dysfunction) who:

* Have stable Class I - III New York Heart Association (NYHA) classification for chronic heart failure
* Have not been hospitalised for an exacerbation of their heart failure in the 6 weeks prior to screening
* Are able to communicate in English (both verbally and in writing)

Exclusion Criteria:

Any patients who have:

* Any severe neuro-psychological or neuro-cognitive conditions that would confound outcome assessment
* NYHA Class IV classification for chronic heart failure receiving end of life care, or other life-threatening condition

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult males and females with suspected Heart Failure with Preserved Ejection fraction
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Morbidity | 1 year from recruitment
  Episodes of diseases
Mortality | 1 year from recruitment
  Confirmed death during follow-up

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire | Baseline, 6 & 12 months
  Heart failure specific quality of life over time (transformed total score 0 - 100); higher scores indicate better quality of life. 5 point change considered clinically relevant.
6 Minute Walk Test | baseline to 6 & 12 months
  physical function changes over time
Montreal Cognitive Assessment (MOCA) | baseline to 6 & 12 months
  cognitive function over time

CONTACTS AND LOCATIONS:
Overall Officials: Christi Deaton, PhD,RN, Principal Investigator — Cambridge University Hospitals NHS FT
Locations (1):
- Cambridge University Hospital NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Austin R, Khair E, Blakeman T, Hossain MZ, Sowden E, Chew-Graham C, Forsyth F, Deaton C; Optimise HFpEF Investigators; Optimise HFpEF Investigators. Diagnosing and managing patients with heart failure with preserved ejection fraction: a consensus survey. BMJ Open. 2024 Dec 20;14(12):e092993. doi: 10.1136/bmjopen-2024-092993. PMID 39806710
- [Derived] Hossain MZ, Chew-Graham CA, Sowden E, Blakeman T, Wellwood I, Tierney S, Deaton C. Challenges in the management of people with heart failure with preserved ejection fraction (HFpEF) in primary care: A qualitative study of general practitioner perspectives. Chronic Illn. 2022 Jun;18(2):410-425. doi: 10.1177/1742395320983871. Epub 2021 Jan 5. PMID 33401942
- See also: Study website — https://www.optimisehfpef.phpc.cam.ac.uk/